CLINICAL TRIAL: NCT02960828
Title: Focal Subthreshold Laser Treatment for Macular Drusen
Brief Title: "Stop Early Age-related Macular Degeneration (AMD) From Vision Loss Eternally" Study
Acronym: SAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyu Hyung Park, Professor, Chief of department of Ophthalmology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1508/312-004
Record Dates: First submitted 2016-06-30; First posted 2016-11-10 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Age-Related Macular Degeneration; Retinal Drusen
MeSH Terms: conditions — Macular Degeneration; Retinal Drusen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention-"Device:_Laser" (Experimental): * Subthreshold focal photocoagulation
  * Intravitreal Anti-vascular endothelial growth factor (Anti-VEGF) injection
  Interventions: Procedure: Subthreshold Laser Photocoagulation; Drug: intravitreal Anti-VEGF injection; Device: Subthreshold Laser
- Control (No Intervention): Contralateral eye

INTERVENTIONS:
Procedure: Subthreshold Laser Photocoagulation — Selective Subthreshold Laser Photocoagulation is applied to the periphery of high-risk macular drusen
  Arms: Intervention-"Device:_Laser"
Drug: intravitreal Anti-VEGF injection — To prevent choroidal neovascularization, intravitreal Anti-VEGF injection is done on a 3 month interval up to 1 year.
  Arms: Intervention-"Device:_Laser"
Device: Subthreshold Laser
  Arms: Intervention-"Device:_Laser"

SUMMARY:
This study aims to validate the efficacy and safety of subthreshold laser photocoagulation on high-risk macular drusen in early age-related macular degeneration which has a high risk of conversion to exudative AMD.

DETAILED DESCRIPTION:
SAVE Study (Stop Early Age-related Macular Degeneration form Vision Loss Eternally)

ELIGIBILITY:
Inclusion Criteria:

* Drusen in both eyes examined under fundoscopy
* At least one of the eyes must have high-risk soft drusen
* BCVA below ETDRS 83 letters
* Patient with consent to participate

Exclusion Criteria:

* Prior diagnosis with choroidal neovascularization
* Exudative AMD in at least one eye
* If the patient has only one visually effective eye (last eye)
* Other macula or retinal diseases than age-related macular degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in drusen size | 3 month interval

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 3 months interval
  ETDRS and Snellen visual acuity measurement
Change in drusen distribution | 3 month interval
Change in autofluorescence | 3 month interval
Choroidal Neovascularization | 3 months interval
Contrast Sensitivity | 3 months interval
  Contrast Sensitivity Test

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyung Park, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyunggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided